CLINICAL TRIAL: NCT06313957
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of LUCAR-20SP, an Allogenic Chimeric Antigen Receptor(CAR)-T Cell Therapy Targeting CD20 in Subjects With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: A Study of LUCAR-20SP in Subjects With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry); Beijing Boren Hospital (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2302-0001
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Relapsed B-cell Non-Hodgkin Lymphoma; Refractory B-cell Non-Hodgkin Lymphoma
Keywords: Relapsed B-cell non-Hodgkin lymphoma; Refractory B-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Each subject will receive LUCAR-20SP cells (Experimental): Chimeric antigen receptor T cells LUCAR-20SP cells
  Interventions: Biological: LUCAR-20SP cells

INTERVENTIONS:
Biological: LUCAR-20SP cells — Prior to infusion of the LUCAR-20SP, subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine.

SUMMARY:
This is a prospective, single-arm, open-label, exploratory clinical study of LUCAR-20SP in adult subjects with relapsed/refractory B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label exploratory clinical study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor efficacy profiles of LUCAR-20SP, an allogenic CAR-T cell therapy in subjects with relapsed/refractory B-cell non-Hodgkin lymphoma. Patients who meet the eligibility criteria will receive LUCAR-20SP infusion. The study will include the following sequential stages: screening, pre-treatment (lymphodepleting chemotherapy), treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in clinical research;
* Age ≥18 years old;
* Eastern Cooperative Oncology Group (ECOG) score 0-1;
* Histologically confirmed large B-cell lymphoma, follicular lymphoma, mantle cell lymphoma, histologically indolent lymphoma to diffuse large B-cell lymphoma; CD20 positive;
* At least one measurable tumor lesion according to the Lugano 2014.
* Expected survival ≥3 months;
* Clinical laboratory values in the screening period meet criteria.
* Effective contraception.

Exclusion Criteria:

* Prior antitumor therapy with insufficient washout period.
* Previous treatment with allogeneic cell and gene therapy (such as CAR-T); Except subjects with evidence that previous allogeneic cell and gene therapy products (such as CAR-positive T cells and CAR transgenes) in the subject have been below the lower limit of detection;
* Previously received allogeneic hematopoietic stem cell transplantation;
* Previously received gene therapy;
* Donor specific antibody (DSA) positive subjects will be excluded;
* Severe underlying diseases;
* Hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C virus ribonucleic acid (HCV RNA) or human immunodeficiency virus antibody (HIV-Ab) positive;
* Presence of other serious pre-existing medical conditions that may limit patient participation in the study. Any condition that, in the investigator's judgment, will make the subject unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate | Minimum 2 years after LUCAR-20SP infusion (Day 1)
  DLT refers to a drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose.
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | Minimum 2 years after LUCAR-20SP infusion (Day 1)
  An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment.
Recommended Phase 2 Dose (RP2D) regimen finding | Minimum 2 years after LUCAR-20SP infusion (Day 1)
  RP2D established through accelerated titration design (ATD) and Bayesian Optimal Interval (BOIN) design.
Pharmacokinetics in peripheral blood | Minimum 2 years after LUCAR-20SP infusion (Day 1)
  CAR transgene levels in peripheral blood after LUCAR-20SP infusion. CAR positive T cells levels in bone marrow after LUCAR-20SP infusion.
Pharmacokinetics in bone marrow | Minimum 2 years after LUCAR-20SP infusion (Day 1)
  CAR positive T cells levels in bone marrow after LUCAR-20SP infusion. CAR transgene levels in bone marrow after LUCAR-20SP infusion.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) after administration | Minimum 2 years after LUCAR-20SP infusion (Day 1)
  ORR is defined as the proportion of subjects who achieve complete response (CR) or partial response (PR) after treatment via LUCAR-20SP cell infusion, and the objective tumor response rate will be calculated for patients with measurable disease per the Lugano Classification for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma (Lugano 2014)
Time to Response (TTR) after administration | Minimum 2 years after LUCAR-20SP infusion (Day 1)
  TTR is defined as the time from the date of first infusion of LUCAR-20SP to the date of the first response evaluation of the subject who has met all criteria for PR or better.
Duration of Remission (DoR) after administration | Minimum 2 years after LUCAR-20SP infusion (Day 1)
  DoR is defined as the time from the first documentation of remission (PR or better) to the first documented disease progression evidence (according to Lugano 2014) of the responders (who achieve PR or better response).
Progression-free Survival (PFS) after administration | Minimum 2 years after LUCAR-20SP infusion (Day 1)]
  PFS is defined as the time from the date of first infusion of the LUCAR-20SP to the first documented disease progression (according to Lugano 2014) or death (due to any cause), whichever occurs first.
Overall Survival (OS) after administration | Minimum 2 years after LUCAR-20SP infusion (Day 1)]
  OS is defined as the time from the date of first infusion of LUCAR-20SP to death of the subject.
Incidence of anti-LUCAR-20SP antibody | Minimum 2 years after LUCAR-20SP infusion (Day 1)
  The incidence of anti-LUCAR-20SP antibody in patients who received LUCAR-20SP infusion.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing GoBroad Boren Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No